CLINICAL TRIAL: NCT06452186
Title: Toward Restoration of Normative Postural Control and Stability Using Neural Control of Powered Prosthetic Ankles
Brief Title: Restoration of Normative Postural Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, He Huang, Professor, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 26076
Record Dates: First submitted 2024-01-29; First posted 2024-06-11 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: powered ankle prosthesis; direct EMG control; balance; cognitive load; muscle synergy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Two groups amputees go through the same training procedure with different prostheses. Their functionality will be compared before and the after the training.
Who Masked: Outcomes Assessor
Masking Description: The PT, who evaluates the participants, is blinded for their previous training experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- dEMG group (Experimental): Patients go through the training procedure with the direct EMG controlled powered prosthetic ankle.
  Interventions: Device: direct EMG controlled prosthetic ankle; Behavioral: PT guided prosthetic training
- Passive group (Active Comparator): Patients go through the training procedure with their own passive prosthetic ankles
  Interventions: Behavioral: PT guided prosthetic training

INTERVENTIONS:
Device: direct EMG controlled prosthetic ankle — Patients are trained to use the powered prosthetic ankles
  Arms: dEMG group
Behavioral: PT guided prosthetic training — Amputees are trained to use prosthetic ankles

SUMMARY:
The objective of this proposal is to investigate the effects of training to use direct electromyographic (dEMG) control of a powered prosthetic ankle on transtibial amputees'.

The aimed questions to answer:

1. whether dEMG control will improve balance and postural stability of amputees,
2. whether dEMG control will lead to more natural neuromuscular control and coordination, 3) whether dEMG control will reduce cognitive processes.

Participants will go through PT guided training on using dEMG controlled prosthetic ankles and are evaluated for their capability on functional tasks.

The results will be compared with a comparison group, which goes through the same training but with their everyday passive prostheses on balance capability, neuromuscular coordination, and cognitive load during locomotion.

DETAILED DESCRIPTION:
Lab Visit Experience for Participants with lower limb amputation:

* Number of Lab Visits: 15 visits. Clinicians may recommend skipping some of the visits or tasks based on clinical evaluation and status of the participants.
* Length of Lab Visit: three hours maximum

  1. First visit: the purpose of the first visit is to conduct consent and conduct measurements to decide walking speed and ABC (amputee balance confidence) score.
  2. Second visit: this visit is to ensure that the amputees' own socket system can be integrated into the powered prosthetic leg and validate the effectiveness of the EMG interface.
  3. Third and fourth visits: baseline evaluation with powered prosthesis and passive prosthesis. Each participant will finish the two visits. One of the visits is dedicated to their own passive prosthesis and the other visit is for the powered prosthesis. The sequence of the evaluation is randomized. The tasks conducted in the two visits are generally identical. The only difference is that one of the visits uses the participants' everyday prosthetic foot and the other uses the powered prosthetic ankle
  4. Fifth and sixth visits: these visits are dedicated to have the participants trained to regain muscle coordination, which is critical to use the powered prosthetic ankle. All the participants will go through these trainings. Based on whether the participants are selected as the powered prosthetic group (Group A) or the passive group (Group B), the participants will finish this training with the powered prosthetic leg or a passive prosthetic leg.
  5. Seven - eleventh visits: These visits are designed to give participants needed training, so participants are able to integrate the action of the powered prosthetic ankle with their full body motion for various tasks. To ensure that contribution of the training procedure to the performance changes are considered, all the participants will go through the training with the prostheses aligned with their group.
  6. Twelfth-thirteenth visit (duplicate of Third and fourth visit). These visits are used to evaluate the impact of the training program on the performance of the participants to conduct tasks which are not included in the training procedure. Each participant will conduct the task with both passive and powered prosthetic legs on different days.
  7. Fourteenth-fifteenth visits (duplicate of Third and fourth visit). These visits are used to understand the long term effects of the training program on the participants. These visits will be conducted three months after the 13th visits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* unilateral bower limb amputee
* K-level 2 or higher (who are frequent prosthesis users and may benefit from the proposed prosthesis training and use of dEMG controlled powered prosthesis)
* Amputation occurred over 2 years ago
* At least 1 year of experience using their prosthetic leg
* Has used the current socket for at least 6 months without a significant skin issue or major modification
* Are willing to come to NC State University's Centennial Campus to participate in research and be photographed while doing research activities

Exclusion Criteria:

* Have a very short residual shank (the length of the residual limb is ≤15% of the length of intact limb)
* Cannot perform functional ambulation in the community on a daily basis without assistive devices
* Cognitive or visual impairment that affects the participant's ability to provide informed consent or to follow simple instructions during the experiments
* Congenital amputees
* Amputees who use powered prosthetic ankles
* Weight more than 300lbs
* Pregnant Person
* Allergic to latex, which is often contained in medical tapes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
aCOM, anticipatory Center of Mass Excursion when the expected disturbance is introduced | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  This measurement is to quantify the movement of the COM at the time when the disturbance is introduced and represents an important element of the capability of the participants to conduct anticipatory. Higher value indicates better capacity to conduct anticipatory postural control.

SECONDARY OUTCOMES:
Frequency of stepping responses | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  Number of amputees to conduct steps to recover from disturbance divided by total number of disturbance, which they experienced.
Zero-time-lag cross correlation coefficients for bilateral ankle torque | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  Torque in the anterior-posterior direction. This outcome quantify the symmetry between the prosthetic ankle and the unaffected ankle when the participants try to maintain balance under expected disturbance
Prosthesis Embodiment Scale | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  The Prosthesis Embodiment Scale for Lower Limb Amputees (PEmbS-LLA) measures amputees' feeling of ownership, sense of agency, and anatomical plausibility of a lower limb prosthetic device. This scale has been tested on lower limb amputees using daily prescribed prosthesis (not neurally controlled) with established validity and reliability. The score range is -3~3 and high value indicates better embodiment.
Average muscle modules structure correlation | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  Correlation coefficient of muscle modules structures identified using nonnegative matrix factorization (NNMF) during a voluntary postural sway task. This measure is used to determine whether muscle modules employed between populations are meaningfully similar.
Scores from Amputee Mobility Predictor (AMP) Test | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  Clinical balance outcomes used to measure the capacity of participants to conduct functional tasks, which are related to balance. The score ranges from 0-47. Higher values indicate better performance.
Scores from MiniBES Test (Balance Evaluation Systems Test ) | Pre-training (before the training starts), Post-training (immediately after the training), and follow-up evaluation (one month) with both passive and dEMG devices
  Clinical balance outcomes used to measure the capacity of participants to conduct functional tasks, which are related to balance. The score ranges from 0 to 28. The higher value indicates better balance capability

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — NC State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

DOCUMENTS (2):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT06452186/Prot_000.pdf
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT06452186/ICF_001.pdf